CLINICAL TRIAL: NCT01144728
Title: AMIT Study - Amaryl M Initiation and Titration Study
Brief Title: Initiation and Titration of Amaryl
Acronym: AMIT KZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLMET_L_04718; U1111-1116-9956 (Other: UTN)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin

ARMS (1):
- Single arm Glimepiride+metformin (Experimental): Start and titration based on FBG and tolerance. Titration should be achieved within maximum 4 weeks.
  Interventions: Drug: GLIMEPIRIDE + METFORMIN

INTERVENTIONS:
Drug: GLIMEPIRIDE + METFORMIN — Pharmaceutical form: Tablet Route of administration: oral Dose regimen : fixed dose combination of glimepiride / metformin: 1/250, 2/500

SUMMARY:
Primary Objective:

* To describe the conditions of initiation and titration of Amaryl M, according to previous treatment:
* initial dose
* titration scheme
* efficacy after 4 months assessed by HbA1C
* tolerability (number and severity of hypoglycaemia)

Secondary Objective:

* Fasting Plasma Glucose
* Weight evolution

ELIGIBILITY:
Inclusion criteria:

* Patients with Type 2 diabetes who have been treated with a stable dose (any dose) of :
* sulfonylurea monotherapy or
* metformin monotherapy or
* free combination of glimepiride and metformin with a stable dose (any dose)
* Body Mass Index (BMI) between 20 and 40 kg/m2
* HbA1c superior or egal to 7.5%
* FPG superior or egal 7 mmol/l

Exclusion criteria:

* Secondary or insulin-dependant diabetes
* Any severe chronic disease (hepatic, renal impairments)
* History of major cardiovascular event in the last 6 months
* Acute conditions with the potential to alter renal function such as: dehydratation, severe infection, shock, IV administration of iodinated contrast agents
* Allergy to sulfonylurea, metformin
* Drug or alcohol abuse
* Pregnancy, lactation

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Glycolysated Haemoglobin (HbA1c) | From baseline to Month 4
Patients With Glycosylated Haemoglobin (HbA1c) Value < 7% | Month 4
Evolution of Fasting Plasma Glucose (FPG) | From baseline to Months 4

SECONDARY OUTCOMES:
Post Prandial Plasma Glucose (PPPG) | Month 4
Number of patients for each start dose | At baseline
Number of patients with different final doses | Month 4
Rate of Symptomatic Hypoglycemia | During treatment period (4 months)
Change in Weight | Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Almaty, Kazakhstan